CLINICAL TRIAL: NCT07129083
Title: Exploring Predictors of Quality of Life in Older Adults With End-Stage Kidney Disease Receiving In-Center Hemodialysis: A Cross-Sectional Analysis of Sociodemographic, Dialysis-specific, Biopsychosocial, and Activity-Related Factors
Brief Title: Exploring Predictors of Quality of Life in Older Adults With End-Stage Kidney Disease Receiving In-Center Hemodialysis
Acronym: B670201837264
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-11716
Record Dates: First submitted 2025-07-18; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: End Stage Renal Failure, Hemodialysis
Keywords: End-stage Kidney Disease; Hemodialysis; Quality of Life; Older Adults
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older adults receiving in-center hemodialysis: Adults aged 65 years and older undergoing maintenance in-center hemodialysis at four hospitals in Flanders, Belgium. Participants completed structured assessments covering overall quality of life, health-related quality of life, clinical, functional, psychological, and sociodemographic variables.
  Interventions: Other: Structured assessment interview

INTERVENTIONS:
Other: Structured assessment interview — Participants completed a structured, in-person assessment conducted during one to three dialysis sessions. The assessment included validated instruments to measure overall quality of life (ACSA), health-related quality of life (EQ-5D-3L, EORTC QLQ-C30, QLQ-MY20), and various clinical, psychological, functional, and sociodemographic factors.

SUMMARY:
This cross-sectional observational study investigates the overall quality of life (QoL) in adults aged 65 and older receiving in-center hemodialysis. While health-related quality of life (HRQoL) is commonly used in nephrology, it may not fully reflect what matters most to older patients. Using the Amnestic Comparative Self-Assessment (ACSA) as the primary measure, this study explores key determinants of QoL and examines how it relates to existing HRQoL tools (EQ-5D-3L, EORTC QLQ-C30, QLQ-MY20). Data are collected from four hospitals in Flanders, Belgium, using psychosocial (geriatric) assessments. Statistical analysis includes regression and cluster methods to identify predictors and patient subgroups. Results aim to inform more patient-centered care and improve QoL measurement in dialysis research.

DETAILED DESCRIPTION:
The global prevalence of end-stage kidney disease (ESKD) is steadily rising, with older adults representing the fastest-growing demographic in this patient population. In Europe, individuals aged 65 and older now account for over 52% of all incident ESKD cases. The primary treatment modality, in-center hemodialysis (ICHD), although life-sustaining, imposes a considerable treatment burden. This burden, when combined with the inherent symptom load of advanced kidney disease, often leads to a significant reduction in patients' overall well-being.

Compared to their younger counterparts, older adults on dialysis experience more complex clinical trajectories, characterized by multi-morbidity, increased frailty, and psychosocial vulnerability. Moreover, this population often faces challenges in adhering to the demanding schedules and lifestyle restrictions associated with dialysis. These factors collectively contribute to a reduction in overall quality of life (QoL), which patients often prioritize even over life expectancy.

Numerous studies have demonstrated that many older dialysis patients are willing to trade significant lengths of life expectancy, up to nine years in some cases, in exchange for better QoL. Despite this, QoL remains a vastly underutilized metric in nephrology clinical research. Only a small fraction of randomized controlled trials include QoL as an outcome measure, and even fewer consider it as a primary endpoint.

Health-Related Quality of Life (HRQoL), a narrower construct within the broader domain of QoL, is often used as a proxy for evaluating the well-being of patients. However, HRQoL tools may not fully capture what matters most to patients, especially during major life transitions such as dialysis initiation. Furthermore, differences in HRQoL instruments can produce inconsistent evaluations of patient outcomes and influence the estimation of quality-adjusted life years (QALYs), potentially skewing health policy decisions.

In light of these concerns, there is a need to examine overall QoL among older adults receiving dialysis, moving beyond standard HRQoL assessments to capture a more holistic and patient-centered understanding of life quality in this vulnerable population.

This study aims to:

* Identify the key determinants of overall QoL in older adults undergoing ICHD.
* Examine how overall QoL relates to existing HRQoL measures.
* Evaluate whether existing HRQoL instruments adequately capture domains that are meaningful to this population.
* Explore natural groupings (clusters) of patients based on QoL and associated variables to inform future patient-centered interventions.

Study Design This is a cross-sectional, observational study reported in accordance with the Strengthening The Reporting of Observational Studies in Epidemiology (STROBE) guidelines. The study involves quantitative data collection through a structured assessment set administered face-to-face during dialysis sessions.

Participants are recruited from four hospitals in the Flanders region of Belgium between January and April 2018. Hospitals are selected to ensure a representative sample across urban, rural, academic, and regional settings.

Eligibility criteria include:

Age ≥65 years Receiving ICHD Able to provide informed consent Sufficient cognitive and language capacity to complete the questionnaire in Dutch

Exclusion criteria include:

Receiving dialysis due to an acute hospital admission Diagnosed with severe psychiatric or cognitive disorders (e.g., dementia) as documented in the medical record

Data Collection and Outcome Measures A total of 95 variables are assessed across multiple domains, guided by the International Classification of Functioning, Disability and Health (ICF) framework. Assessments are conducted during one to three consecutive dialysis sessions, depending on each participant's physical and cognitive condition. Each session lasts approximately 45 minutes.

An independent researcher with no clinical ties to the patient or dialysis unit conducts all interviews to reduce bias and minimize socially desirable responses.

Primary Outcome Measure Amnestic Comparative Self-Assessment (ACSA): A self-anchoring QoL rating scale ranging from -5 (worst period of life) to +5 (best period), based on the individual's life experiences. Participants reflect on the most positive and negative periods of their life and rate their current quality of life relative to these anchors. This tool allows for a highly individualized and sensitive measure of overall QoL.

Secondary Measures (Independent Variables) Sociodemographic Variables: Age, sex, education level, marital status, living situation Dialysis-Related Variables: Duration of dialysis, comorbidity index, dialysis adequacy Comprehensive Geriatric Assessment (CGA): Functional, psychological, and social domains including Fall Risk: STRATIFY scale, Psychological Measures: Geriatric Depression Scale (GDS-4), Nutritional Status: Nutritional Risk Screening (NRS-2002) Frailty Assessment: Groningen Frailty Indicator (GFI) Functional Status: Brussels Integrated Activity Scale (BIA) - measuring basic, instrumental, and advanced ADLs

HRQoL Instruments:

EuroQol 5-Dimension 3-Level Questionnaire (EQ-5D-3L) European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) EORTC QLQ-Myeloma Module (QLQ-MY20)

Statistical Analysis

All data are analyzed using SPSS (version 29.0.2.0). Missing values are handled using listwise deletion per questionnaire. The analysis is carried out in four stages:

1. Descriptive Statistics: Means and standard deviations for normally distributed variables, medians and interquartile ranges for non-normal distributions. Normality assessed via Shapiro-Wilk test.
2. Univariate Analyses:

   Mann-Whitney U test for dichotomous variables Kruskal-Wallis test for categorical variables with more than two groups Spearman's correlation for continuous and ordinal variables
3. Multivariate Regression: Variables significantly associated with ACSA scores in univariate analysis are entered into a stepwise linear regression model to identify independent predictors of QoL.
4. Cluster Analysis: Hierarchical clustering (Ward's method) is used to determine optimal grouping, followed by K-means clustering to explore patterns of QoL across patient subgroups.

Ethical Considerations This study was reviewed and approved by the Ethical Committee of Ghent University Hospital (B670201837264). All participants are fully informed of the study's purpose and procedures and provided both written and verbal informed consent. The study complies with the Declaration of Helsinki on ethical principles for medical research involving human subjects.

Significance and Expected Outcomes

This study offers an exploration of overall QoL in older adults receiving hemodialysis. By using the ACSA alongside commonly used HRQoL instruments and a wide range of biopsychosocial variables, the findings will help:

1. Clarify which factors most strongly influence QoL in this population
2. Reveal potential mismatches between standardized HRQoL measures and patients' lived experiences
3. Inform future intervention design focused on improving well-being, not just clinical outcomes
4. Provide empirical evidence to guide the choice of QoL instruments in research and policy evaluation, including cost-effectiveness studies

Ultimately, the study is expected to contribute to more patient-centered care models and improve the integration of QoL measures into nephrology research and clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Receiving maintenance in-center hemodialysis (ICHD)
* Able to provide informed consent
* Sufficient cognitive capacity to understand and answer study questions
* Fluent in Dutch (able to complete assessments in Dutch)

Exclusion Criteria:

* Receiving ICHD due to an acute hospital admission (not chronic treatment)
* Documented diagnosis of severe psychiatric illness or severe cognitive impairment (e.g., dementia)
* Unable to understand or respond adequately to the questionnaire

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older adults with end-stage kidney disease undergoing maintenance in-center hemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Quality of Life - Amnestic Comparative Self-Assessment (ACSA) | Baseline
  A self-anchoring Quality of Life scale ranging from -5 (worst time in life) to +5 (best time in life). Participants reflect on their personal best and worst life periods and rate their current QoL accordingly.

SECONDARY OUTCOMES:
Age | Baseline
  Age (in years)
Marital status | Baseline
  Marital status (single, married, widowed)
Living situation | Baseline
  Living situation (independently alone, independently with family, in a care facility)
(Grand)children | Baseline
  (Grand)children (yes/no, number of children and grandchildren)
Dialysis vintage | Baseline
  Dialysis vintage up to baseline measure (in months)
Hospital admissions | Baseline
  Hospital admissions (amount in the last year)
Risk of falls | Baseline
  St. Thomas's Risk Assessment Tool in Falling Elderly Inpatients (STRATIFY); minimum score = 0, maximum score = 5; higher score indicates a higher risk of falling
Risk of dementia | Baseline
  Risk of dementia using Mini-Cog (full name); minimum score = 0, maximum score = 5; lower score is higher risk of dementia
Nutritional risk | Baseline
  Nutritional risk using the Nutritional Risk Screening 2002 (NRS-2002); minimum score = 0, maximum score = 7; lower score (<3) = lower nutritional risk
Experienced level of pain | Baseline
  Pain, measured using a VAS-scale (from 0= no pain, to 9= worst pain imaginable)
Vision impairment | Baseline
  Potential vision impairment, measured using two questions: 1. Do you have vision problems?; 2. Do you wear glasses?
Hearing impairment | Baseline
  Potential hearing impairment, measured using two questions: 1. Do you have hearing problems?; 2. Do you use hearing aids?
Continence problems | Baseline
  Potential continence problems, measured using two questions: 1. Do you have problems with continence?; 2. Do you use continence material?
Frailty | Baseline
  The Groningen Frailty Indicator (GFI), a multidimensional frailty measure; minimum score = 0, maximum score = 15; Higher score (≥4) implies (higher levels of) frailty
Activity | Baseline
  Brussels Integrated Activity Scale (BIA), measuring basic-, instrumental-, and advanced activities of daily living; Minimum score = 0 (completely dependent in all activities), maximum score = 54 (completely independent in all activities); Higher score = better functional status / greater independence
Health-Related Quality of Life: EQ-5D-3L | Baseline
  Health-related quality of life assessed using the EuroQol 5-Dimension 3-Level questionnaire (EQ-5D-3L); includes 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), rated at 3 levels (1= no problems, 2= some problems, 3= unable to/extreme problems). These can be converted into a utility score ranging from +- -0.59 to 1.00 (higher = better health). The EQ5D also includes a VAS-scale, where self-perceived health is rated from 0 (worst) to 100 (best)
Health-Related Quality of Life using the EORTC QLQ-C30 | Baseline
  The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30) measures health-related quality of life through 5 functional, 9 symptom, and 1 global health status scale; minimum score = 0, maximum score = 100 (for functional scales, higher is better; for symptom scales, lower is better)
Health-Related Quality of Life: EORTC QLQ-MY20 | Baseline
  The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Multiple Myeloma Module (EORTC QLQ-MY20) measures functioning and symptoms; minimum scores = 0; maximum scores = 100; for all scales, a higher score = worse outcomes (unlike the QLQ-C30 where functional scales mean better functioning)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Van d Van de Velde, Doctorate, Principal Investigator — University Ghent; Wim Van Biesen, Doctorate, MD, Study Director — University Ghent; Patricia De Vriendt, Doctorate, Study Chair — University Ghent
Locations (1):
- Ghent University Hospital, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No
Not applicable. There is no plan to share individual participant data.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT07129083/Prot_SAP_000.pdf